CLINICAL TRIAL: NCT01515280
Title: Supplementary Study of Hull Airway Reflux Questionnaire Scores Before and After Treatment Study: A Multicentre, Double-Blind, Placebo-Controlled, Pivotal Study of the Efficacy and Safety of Oral Theobromine in the Management of Cough."
Brief Title: Hull Airway Reflux Questionnaire Scores Following Cough Treatment
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 11112011
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Cough
Keywords: chronic cough
MeSH Terms: conditions — Cough; Chronic Cough

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic cough: Patients taking part in supplementary study must be randomised to main study which includes a placebo arm and treatment arm

SUMMARY:
The aim of this study is to have those patients taking part in the Clinical trial-: A Multicentre, Double-Blind, Placebo-Controlled, Pivotal Study of the Efficacy and Safety of Oral Theobromine in the Management of Cough. Complete the Hull Airway Reflux Questionnaire (HARQ) at randomisation and repeat the questionnaire at the end of the 14 day treatment period. The investigators hope to demonstrate a clinically significant change in HARQ scores of at least 16 points from before and after treatment. Furthermore the investigators would hope to show a significantly improved HARQ score in patients on the BC036 arm of the study compared to the placebo arm.

ELIGIBILITY:
Inclusion Criteria:

1. Male/females meeting eligibility criteria for study: - A Multi-centre, Double-Blind, Placebo-Controlled, Pivotal Study of the Efficacy and Safety of Oral BC1036 in the Management of Cough.
2. Willing and able to comply with study procedures
3. Able to provide written informed consent to participate

Exclusion Criteria:

1. Any subject meeting any exclusion criteria on the study "A Multi-centre, Double-Blind, Placebo-Controlled, Pivotal Study of the Efficacy and Safety of Oral BC1036 in the Management of Cough." Will be excluded from this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients attending chronic cough clinics
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Hull Airway Reflux Questionnaire score | baseline and 2 weeks later
  The primary objective is to evaluate the effectiveness of HARQ in measuring a clinically significant change in HARQ score from baseline following 14 days treatment.

SECONDARY OUTCOMES:
HARQ SCORES | baseline and 14 days
  The Key secondary endpoint will be to evaluate ability of HARQ in demonstrating a clinically significant change in score from baseline in the BC036 arm compared to Placebo arm of main study.

CONTACTS AND LOCATIONS:
Overall Officials: Alyn H Morice, MD, Mphil, Principal Investigator — Hull and EastYorkshire NHS Trust
Locations (1):
- Hull and East Yorkshire Hospitals Trust, Cottingham, East Riding Of Yorkshire, United Kingdom

REFERENCES:
- [Result] Morice AH, McGarvey L, Pavord ID, Higgins B, Chung KF, Birring SS. Theobromine for the treatment of persistent cough: a randomised, multicentre, double-blind, placebo-controlled clinical trial. J Thorac Dis. 2017 Jul;9(7):1864-1872. doi: 10.21037/jtd.2017.06.18. PMID 28839984
- See also: Publication Link — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5542984/